CLINICAL TRIAL: NCT01437124
Title: Measurement of Metal Ion Levels and Chromosome Abnormalities in Ceramic on Metal Total Hip Arthroplasty in Vivo
Brief Title: Metal Ions in Ceramic on Metal Total Hip Arthroplasty
Acronym: COM
Status: Completed | Type: Observational
Sponsor: Hussain Kazi (Other)
Responsible Party: Sponsor-Investigator, Hussain Kazi, Specialist Registrar, Trauma and Orthopaedics, Wirral University Teaching Hospital NHS Trust
Organization: Wirral University Teaching Hospital NHS Trust (Other)
Other Study IDs: 960558216
Record Dates: First submitted 2011-09-16; First posted 2011-09-20 (Estimated); Results first posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-04

CONDITIONS: Osteoarthritis; Avascular Necrosis; Rheumatoid Arthritis; Developmental Dysplasia of the Hip
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis; Arthritis, Rheumatoid; Developmental Dysplasia of the Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ceramic on metal THA: Those who have received a ceramic on metal total hip replacement

SUMMARY:
The investigators aim to measure the blood levels of certain metals in a group of patients all of whom have had a ceramic on metal total hip replacement. This new bearing surface (joint) is relatively new and the investigators are currently following up the largest cohort in the world. Clinical results are currently excellent at 2 years in all patients, however the investigators are mindful of the lessons learned from the high failure rate of several designs of metal on metal hip replacements as well as several in vitro reports and one in vivo case report of elevated metal levels in this particular implant. The investigators feel it is important to measure the metal ion levels in our group to ascertain and compare these with reference standards. Once performed the investigators can relate ion levels to function and x ray changes and provide useful longterm data to the patients and the wider medical community as to whether this bearing surface is safe in the long term or whether it's use should be abandoned. This is useful as there are numerous groups implanting this device in the UK and in addition it has just been awarded FDA approval in the USA - its use is likely to flourish.

DETAILED DESCRIPTION:
PURPOSE & DESIGN:

The investigators are currently following up a cohort of patients all of whom have had a metal on ceramic total hip arthroplasty.

This new bearing couple has been approved for use in the UK for some time and has recently achieved USA FDA approval.

The attraction of this bearing couple is a low rate of wear with reduced complications associated with ceramic on ceramic bearing such as bearing fracture.

Of recent media attention has been the unacceptably high failure of the DePuy ASR metal on metal hip resurfacing. This metal on metal bearing couple has been associated with increased ion levels and chromosome abnormalities in vivo.

In vitro studies and small in vivo studies have revealed much lower wear, particle numbers and ion levels in ceramic on metal studies than in metal on metal bearing surfaces; however there is no large scale evidence that this is the case.

The investigators currently are following up the largest worldwide series of ceramic on metal bearings and clinical results are excellent. It is important however to obtain hard data on metal ion levels in this population firstly to ensure the long term function and health of this cohort but also to provide a barometer for other surgeons who will be using a prosthesis that as yet has little in the way of long term follow up and data on ion levels in a large cohort.

If the ion levels are unacceptably high then the investigators will need to follow these patients closely and offer revision surgery if there are clinical concerns.

For similar reasons it is important to monitor for chromosomal abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Complete history and physical examination
* Previously performed ceramic on metal total hip replacement
* An understanding of the purpose of the study and signed consent form

Exclusion Criteria:

* Hip arthroplasty other than ceramic on metal bearing
* Mentally infirm / incapacitated
* Incomplete history or physical examination
* Unwillingness to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those who have received a ceramic on metal total hip arthroplasty
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2011-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fintan A Carroll, MBBS, FRCS, Study Director — Consultant Orthopaedic Surgeon; Hussain A Kazi, MBChB,FRCS, Principal Investigator — Specialist Registrar, Trauma & Orthopaedics
Locations (1):
- Wirral University Teaching Hospitals NHS Foundation Trust, Metropolitan Borough of Wirral, Merseyside, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ceramic on Metal THA
Started | 83
Completed | 83
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ceramic on Metal THA
Number analyzed (Participants) | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 73
  >=65 years | 10
Age, Continuous [Mean (Full Range); unit: years] | 58 [42 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 45
Region of Enrollment [Number; unit: participants]
  United Kingdom | 83

OUTCOME MEASURES:

1. Primary Outcome: Cobalt Chromium Levels
Description: Serum cobalt chromium levels post THR
Time Frame: 2 years post THR
Population: metal ion levels
Measure: Mean (95% Confidence Interval); unit: micrograms/dl
Arm/Group | Ceramic on Metal THA
Number analyzed (Participants) | 83
micrograms/dl | 1.06 [0.05 to 7.22]

2. Secondary Outcome: Chromosomal Abnormality
Description: Deviation of karyotype from normal 2 years post THR
Time Frame: 2 years post THR
Population: 24 colour FISH
Measure: Mean (95% Confidence Interval); unit: % chromosomal abberations
Arm/Group | Ceramic on Metal THA
Number analyzed (Participants) | 83
% chromosomal abberations | 0.11 [0 to 0.25]

ADVERSE EVENTS:
Arm/Group | Ceramic on Metal THA
Serious Adverse Events (participants affected / at risk) | 0/83
Other Adverse Events (participants affected / at risk) | 0/83

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No